CLINICAL TRIAL: NCT02896790
Title: From the Model to the Adaptation of a Therapeutic Education Program in Cancer Research: the Case of Renal Cancer Patients Treated by Oral Treatments, Multidisciplinary Approach
Brief Title: From the Model to the Adaptation of a Therapeutic Education Program (TEP) in Cancer Research
Acronym: MODAP
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2014/31
Record Dates: First submitted 2016-06-27; First posted 2016-09-12 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Health Services Research
Keywords: Cancer; Oral Therapy; Compliance; Anthropology; Psychology
MeSH Terms: conditions — Neoplasms; Patient Compliance | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Stage 1: Patients without therapeutic education
  Interventions: Other: Interviews with 2 oncologists and 10 patients
- Stage 2: Patients with therapeutic education
  Interventions: Other: Interviews with 15 patients

INTERVENTIONS:
Other: Interviews with 2 oncologists and 10 patients
  Groups: Stage 1
Other: Interviews with 15 patients
  Groups: Stage 2

SUMMARY:
The use of oral targeted therapies draws new medical management but also new practices for the patients (compliance), their family and the healthcare professionals [1,2]. These therapies have sometimes heavy toxicity: side effects to identify, to treat, and for the patient to learn to manage. This situation underlines the importance of a therapeutic education to accompany this "learning" [3]. Nevertheless, in France, the therapeutic educational programs, built according to the "standards" of the therapeutic education (TE), are still very rare in cancer research [4]. In May 2012, a therapeutic educational program for these patients has been developed in the oncology department of the Teaching Hospital of Bordeaux through a multidisciplinary team. This program, dedicated to metastatic renal cancer patients treated by oral targeted therapies, becomes here an object of research: MODAP (action-research).

DETAILED DESCRIPTION:
At the diagnosis, 25 to 30 % of renal cancer patients present a metastatic disease. The prognosis remains dark in spite of the advent of the targeted therapies from 2007. Actually, the use of oral targeted therapies, most of the time carried out on an outpatient basis (sunitinib in particular), draws new medical management but also new practices for the patients (compliance), their family and the healthcare professionals [1,2].

These therapies have sometimes heavy toxicity: side effects to identify, to treat, and for the patient to learn to manage. This situation underlines the importance of a therapeutic education to accompany this "learning" [3]. Nevertheless, the therapeutic educational programs, built according to the "standards" of the therapeutic education (TE), are still very rare in cancer research [4]: multiplicity of the pathology (a cancer, cancers), multiplicity of the patients' experiences, the difficulty of implementation? In May 2012, in front of the experience told by the patients and the professionals in the context of metastatic renal cancer, the members of the oncology department of the Teaching Hospital of Bordeaux, the therapeutic educational Federation, the Coordination Cancer Centre (3C), an anthropologist, an expert patient and a patient's association developed a therapeutic educational program for these patients [current approval].

This program, built on the model of the TE in France, becomes here an object of research: MODAP (action-research).

ELIGIBILITY:
Inclusion Criteria:

* Age = 18 years old
* Metastatic Renal cancer (carcinoma with clear cells and other subcategories)
* Indication of a first line of treatment of therapy targeted by Sutent ©
* General WHO 0-2 state
* Life expectancy = 12 weeks
* Agree to participate in MODAP (Therapeutic Education)

Exclusion Criteria:

* History of other cancer
* History of severe psychiatric affection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Metastatic Renal cancer
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2015-03-09 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Health quality of life with QLQC30 questionnaire | Three years

SECONDARY OUTCOMES:
Participation rate to the program stages | Two years
  Quantitative data analysis of questionnaires about the health program satisfaction Participation rate to the program stages Attendance to the program stages Management of therapeutic plan : number of rendez-vous changed by the patient or healers
Number of rendez-vous changed by the patient | Two years
Number of rendez-vous changed by the healers | Two years
Number of therapeutic education procedures stages versus the number realized | Two years
Number of calls by nurses | Two years
  Management of therapeutic plan : number of rendez-vous change by the patient or healers, number of therapeutic education procedures stages versus the number realized, number of calls by nurses

CONTACTS AND LOCATIONS:
Overall Officials: Hélène HOARAU, PhD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Hôpital Saint-André, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gross-Goupil M, Escudier B. [Targeted therapies: sequential and combined treatments]. Bull Cancer. 2010;97:65-71. doi: 10.1684/bdc.2010.1071. French. PMID 20418205
- [Background] Hoarau H, Giacomoni C, Etienne G, Fort MP, Mahon FX, Ceccaldi J, Reiffers J, Monnereau A. Expérience quotidienne des patients atteints de LMC traités par voie orale : déterminants des pratiques d'observance ?. Oncologie, 2012, n° 14, p. 609-612.
- [Background] Santucci R, Aatmani AE, Lescoute A, Leveque D, Serra S, Bergerat JP, Beretz L, Herbrecht R. [Potential clinical impact of therapeutic education in patients treated with anticancer drugs]. Bull Cancer. 2011 Feb;98(2):176-81. doi: 10.1684/bdc.2011.1308. French. PMID 21382797
- [Background] Regnier Denois V, Poirson J, Nourissat A, Jacquin JP, Guastalla JP, Chauvin F. Adherence with oral chemotherapy: results from a qualitative study of the behaviour and representations of patients and oncologists. Eur J Cancer Care (Engl). 2011 Jul;20(4):520-7. doi: 10.1111/j.1365-2354.2010.01212.x. Epub 2010 Jul 23. PMID 20649809